CLINICAL TRIAL: NCT00976417
Title: Mechanisms of Action of Adaptive Servoventilation: Ventilatory Control in Heart Failure Patients With Central Sleep Apnoea
Brief Title: Mechanisms of Action of Adaptive Servoventilation
Status: Completed | Type: Observational
Sponsor: ResMed (Industry)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 09/H0708/35
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-11

CONDITIONS: Heart Failure; Sleep Apnea Syndromes
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1. Patients in the control group
- 2. Patients in the intervention group

SUMMARY:
It is known that a significant proportion of patients with heart failure have sleep disordered breathing (SDB). Some of these patients will have Central Sleep Apnoea which is one form of SDB. The SERVE-HF study aims to look at the effect of a breathing support machine, or ventilator called Adaptive Servo-ventilation (ASV) on mortality in heart failure patients with central sleep apnoea. In this related sub-study the investigators want to look at how the ASV machine has its effect. The investigators will be carrying out tests in the laboratory to measure various aspects of the way that breathing is controlled to measure the effect that ASV has on patients.

In addition measurements looking at activity levels will be made using an actiwatch device worn by patients for 14 consecutive days and nights.

Healthy controls will be recruited to all parts of this protocol (ie measurements at baseline and 3 months) to allow comparison of data between patients and controls.

DETAILED DESCRIPTION:
As part of a wider study we are interested in how patients with a failing heart breathe during sleep. It is known that patients with heart failure and central sleep apnoea (a form of breathing difficulty during sleep) have a poorer prognosis. It is likely that this is because this condition places an extra strain on the heart. We want to investigate whether or not treating these breathing problems is of benefit to this group of patients. The proposed study will investigate why a significant proportion of patients with heart failure have central sleep apnoea and how they respond to treatment. We will do this by measuring some of the factors which contribute to how they breathe:

(i) How the brain changes the breathing rate and depth in response to a change in carbon dioxide levels (Chemosensitivity); (ii) How the blood vessels in the brain change in response to a change in carbon dioxide levels (Cerebral Vascular Reactivity); (iii) An overall measure of breathing control called "Loop Gain" (this protocol will only be undertaken in a subgroup of patients who will give specific consent).

These measurements will be carried out in the laboratory in patients taking part in SERVE-HF; a multicentre randomised controlled study of adaptive servoventilation (ASV). ASV is a form of non-invasive ventilation (delivered by a mask worn on the face) shown in previous smaller studies to adequately suppress sleep disordered breathing. The proposed study will allow us to take measurements from patients assigned to both the treatment and control groups; and compare measurements made in both groups at the start of treatment and at three months.

In addition measurements looking at activity levels will be made using an actiwatch device worn by patients for 14 consecutive days and nights. Previously it has been demonstrated that heart failure patients with sleep disordered breathing have lower levels of daytime activity when compared to heart failure patients without sleep disordered breathing. We will investigate the effect of ASV on activity measurements on this patients with sleep disordered breathing.

Healthy controls will be recruited to all parts of this protocol (ie measurements at baseline and 3 months) to allow comparison of data between patients and controls.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Severe Chronic Heart Failure (CHF) with NYHA class III-IV or NYHA class II with at least one hospitalisation for HF within the last 12 months
* Left ventricular ejection fraction (LVEF) <40% by means of echocardiography, radionucleotide angiography, left ventriculography or cardiac MRI documented less than 12 weeks before randomisation
* Diagnosis of sleep disordered breathing SDB (apnoea-hypopnoea-index (AHI >15/h) with ≥ 50% central events and a central AHI ≥ 10/h)
* Clinically stable with no change in medication and no hospitalisation in preceding month
* Optimised medical treatment according to the applicable guidelines
* Able to provide informed consent

Exclusion Criteria:

* Significant chronic obstructive pulmonary disease (COPD) with Forced Expiratory Volume within one second (FEV1) <50%
* Oxygen saturation at rest during the day ≤ 90% at inclusion
* Current use of Positive Airway Pressure (PAP) therapy
* Life expectancy < 1 year for diseases unrelated to chronic heart failure
* Cardiac surgery, Percutaneous coronary intervention (PCI), Myocardial Infarction (MI) or unstable angina within 6 months prior to randomisation
* Implantation of ICD (implanted cardiodefibrillator) or CRT (cardiac resynchronisation therapy) scheduled or within 6 months prior to randomisation
* Transient ischemic attack (TIA) or Stroke within 3 months prior to randomisation
* Primary hemodynamically significant uncorrected valvular heart disease, obstructive or regurgitant, or any valvular disease expected to lead to surgery during the trial
* Acute myocarditis/pericarditis within 6 months prior to randomisation
* Untreated or therapy refractory Restless legs Syndrome (RLS)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients already recruited to the SERVE-HF study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Morrell, PhD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital and Imperial College, London, United Kingdom